CLINICAL TRIAL: NCT04004676
Title: Effect of Ketone Supplementation on Glycogen Replenishment and Time Trial Performance Following Glycogen Lowering Exercise
Brief Title: Ketone Supplementation, Glycogen Replenishment and Time Trial Performance Following Glycogen Lowering Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Professor, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 113713
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Ketonemia; Exercise Performance; Ketosis
Keywords: Ketones; Glycogen replenishment; Exercise Performance
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: This will be a double blind repeated measures cross over study. There will be two treatments involved: cabohydrate-ketone supplements and carbohydrates alone (placebo). Participants will complete the protocol twice and the treatment order will be systematically rotated to avoid any order effect. Design of the study is composed of a glycogen depleting exercise session, followed by 4 hours of recovery/supplementation, and a 20 km cycling time trial. All participants will arrive in a fasted state to the laboratory. a glycogen depleting exercise bout will be done followed by a 4 hour recovery period. during this 4 hours, participants will ingest the corresponding treatment for the first 2 hours. after recovery, they will perform a 20 km cycling time trial.
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded as an individual not involved in the project will assemble and distribute the treatment (drinks) according to a coding system that is kept confidential until the study is completed. Participants will complete the protocol three times and the treatment order will be systematically rotated to avoid any order effect. taste and texture of treatments will be matched and will be distribute in opaque bottles to keep participant blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Active Comparator): isocaloric carbohydrate - only containing drink will be ingested post glycogen lowering exercise, followed by a 20 km time trial intervention
  Interventions: Behavioral: 20 km time trial performance; Behavioral: Glycogen lowering exercise
- Ketone_CHO (Experimental): Ketone - Carbohydrate supplementation will be ingested post glycogen lowering exercise, followed by a 20 km time trial intervention
  Interventions: Behavioral: 20 km time trial performance; Behavioral: Glycogen lowering exercise

INTERVENTIONS:
Behavioral: 20 km time trial performance — 20 km time trial cycling test will be conducted to measure the effect of different drinks on performance time
Behavioral: Glycogen lowering exercise — Glycogen will be lowered using a 10-min warm-up period at a workload of 50% max wattage power output (Wmax). Thereafter, participants will be instructed to cycle 2-min block periods at alternating workloads of 90% and 50% of Wmax, respectively. This will be continued until the participants are no longer able to complete the 2 min at 90% Wmax. That moment will be defined as the time at which the individual is unable to maintain cycling speed at 60 revolutions/min. At that moment the high-intensity block will be reduced to 80% Wmax. Again, athletes will cycle until they are unable to complete a 2-min block at 80% Wmax, after which the high-intensity block will be reduced to 70% Wmax. Finally, participants will be allowed to stop when pedalling speed could not be maintained at 70% Wmax.

SUMMARY:
20 healthy trained males will volunteer to participate in this study. there will be 2 treatments: Carbohydrate- ketone supplementation and carbohydrate alone. The purpose of this study is to evaluate the effect of glucose-ketone supplementation on a 20 km cycling time trial with a 2-hour feeding during a 4-hour recovery period following glycogen depleting exercise.

DETAILED DESCRIPTION:
Carbohydrates (starches & sugars) are important muscle fuel for exercise at moderate to high intensities. Low glycogen content (stored form of carbohydrates in the body) is associated with fatigue. Thus, greater initial glycogen content has been associated with better performance not only in high intensity intermittent sports, but also in prolonged endurance sports. Dose-response studies have determined that ingestion of 1.2 g·kg-1·h-1 of CHO is the appropriate acute recovery dose to optimize glycogen repletion, with no apparent benefit at higher doses. Protein in combination with CHO has also been proposed to enhance glycogen resynthesis when 1 part protein is provided with ~4 parts CHO. Both strategies, optimal CHO intake and CHO in combination with protein for glycogen resynthesis, have resulted in better exercise performance a few hours after a depleting exercise bout. A recent study provided athletes with ketone esters in a drink after glycogen depleting exercise and found that in the presence of high glucose availability, ketone esters increased glycogen stores by 50% compared to a no ketone, high carbohydrate treatment. However, the authors of this study provided a large quantity of carbohydrates intravenously to maintain blood glucose at 10Mm/L. Consequently, it is unknown whether or not ingesting glucose at the optimal dosage would have the same effect. Furthermore, it is unclear whether or not this difference would translate into improved performance in efforts of more moderate duration. Therefore, the purpose of this study is to assess the effect of glucose-ketone supplementation on a 20 km cycling time trial with a 2-hour feeding during a 4-hour recovery period following glycogen depleting exercise.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study you must be a healthy male or female exercise trained individual (at least 1y training experience - at least 3x week), aged 18-40 years.

Exclusion Criteria:

* have not involved been involved in regular exercise (at least 3x week for at least the past year)
* Have symptoms or take medication for respiratory, cardiovascular, metabolic, neuromuscular disease
* Use any medications with side effects of dizziness, lack of motor control, or slowed reaction time
* Are taking part in another research study
* For women, if you are pregnant or become pregnant during the study.
* Have a history of concussion/head injuries.
* Have an excessive alcohol intake (>2 drinks/day)
* Are a smoker

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
20 km cycling time trial | 40 minutes
  participants will ride for 20 km on a stationary bike and time to finish will be measured

SECONDARY OUTCOMES:
Blood insulin | 2 hours
  insulin in blood will be measured using ELISA kits
Blood Lactate | 45 minutes
  blood lactate will be measured using lactate meter
Blood Ketones | 2 hours
  Ketones in blood will be measured using ketone meter

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western Universiy
Locations (1):
- Exercise Nutrition Laboratory (Western University), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No